CLINICAL TRIAL: NCT00425334
Title: A Clinical Safety (Phase II) Increasing Dose Study of MP4 (Hemospan®) in Total Prostatectomy Surgical Patients
Brief Title: Safety Study of Hemospan® in Prostatectomy Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sangart (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 6012
Record Dates: First submitted 2007-01-18; First posted 2007-01-22 (Estimated); Last update posted 2013-08-19 (Estimated); Status verified 2013-08

CONDITIONS: Blood Loss, Surgical; Prostate Cancer; Surgery
Keywords: Blood loss; Ischemia; Hemoglobin; Blood Substitutes; Plasma Expanders
MeSH Terms: conditions — Blood Loss, Surgical; Prostatic Neoplasms; Hemorrhage; Ischemia | interventions — maleimide-polyethylene glycol-modified hemoglobin, MP4; Ringer's Lactate; Ringer's Solution

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Hemospan (MP4OX) (Experimental): 4.3 g/dL MalPEG-Hb solution
  Interventions: Drug: Hemospan (MP4OX)
- Control (Active Comparator): Ringer's lactate
  Interventions: Drug: Ringer's lactate

INTERVENTIONS:
Drug: Hemospan (MP4OX) — 250 mL or 500 mL Hemospan (MP4OX)
  Other Names: MP4OX solution; 4.3 g/dL MalPEG Hb; PEGylated Hb
  Arms: Hemospan (MP4OX)
Drug: Ringer's lactate — 250 mL or 500 mL Ringer's lactate USP
  Other Names: Lactated Ringers; Ringers solution; Hartmann's solution
  Arms: Control

SUMMARY:
This is a progressive dose escalation study designed to evaluate the safety of Hemospan compared to a standard crystalloid solution (Ringer's lactate) in elective surgery patients undergoing total prostatectomy procedures with anticipated blood loss of more than 500 mL. Secondary objectives of this study are to observe possible activity of Hemospan for tissue oxygenation, perfusion and cardiovascular support.

DETAILED DESCRIPTION:
Donor (allogeneic) blood transfusions are often required during and/or after elective surgery to maintain adequate hemoglobin concentration, prevent tissue ischemia (inadequate perfusion), treat hypotension (low blood pressure), and compensate for fluid shifts. Hemospan is a novel hemoglobin-based oxygen carrier and plasma expander specifically developed to perfuse and oxygenate tissue at risk for ischemia and hypoxia (insufficient oxygenation). As a result of the molecular size and oxygen dissociation characteristics, Hemospan selectively off-loads oxygen in tissues predisposed to low oxygen tension.

In preclinical studies Hemospan has been found to be free of significant toxicity in a variety of animal species. These studies have also demonstrated that Hemospan may be ideally suited for this application, and may even perform better than blood in certain situations. Hemospan has been evaluated in three clinical studies, including a 90-patient multi-center Phase II orthopedic surgery trial completed in Sweden in 2005. No serious adverse events attributable to Hemospan have been noted in any of these trials.

Sangart is developing Hemospan as an oxygen-carrying plasma expander and hemodiluent for patients undergoing elective surgical procedures. In the current Phase II study in prostatectomy patients, the administration of Hemospan (Treatment) or Ringer's lactate (Controls) occurs after approximately 250 mL of surgical blood loss has occurred. Study evaluations include clinical observations, subjective symptoms, vital signs, ECG, pulmonary hemodynamics (by TEE), serum chemistry, hematology, urinalysis, renal function, and oxygenation measurements, as well as a safety follow-up assessment at 4-6 weeks after surgery. An independent Data Safety Monitoring Board (DSMB) will review the safety data following completion of each dosing cohort.

ELIGIBILITY:
Inclusion Criteria:

* Adult male ASA class I or II patients over the age of 18 scheduled for elective total prostatectomy surgery with anticipated blood loss greater than 500 mL
* Patients must be in good health (other than the indication for prostatectomy surgery) as determined by medical history, physical examination, clinical laboratory studies and electrocardiogram (ECG)
* At screening (within 2 weeks of the scheduled surgery) the blood chemistry and hematology (Hb, Hct, RBC, WBC, platelets, PT, PTT, plasma fibrinogen, fibrin split products and haptoglobin) must be within the laboratory normal limits
* Patients must test negative for HIV and hepatitis screens
* Patients must sign an Informed Consent Form (see Appendix II) for the study, which has been reviewed and approved by the Institutional Review Board, prior to screening and entry into the study
* Patients must be available within the continental United States for the period of this study, and willing to complete the follow-up at 4-6 weeks
* Patients must be able to understand and read English

Exclusion Criteria:

* Any acute or chronic condition which would limit the patient's ability to complete the study or jeopardize the safety of the patient
* History or clinical manifestations of a significant cardiovascular or pulmonary disorder
* Clinically significant psychiatric disorder requiring active treatment
* History of diabetes requiring active treatment
* History or clinical manifestation of significant renal or hepatic disorder
* History of thyroid disease or clinical symptoms consistent with thyroid disease
* History of bleeding disorder
* History or family history of a hemoglobinopathy
* Patients with contraindications to TEE probe insertion
* Patients who have received any other investigational drugs within 30 days prior to administration of the study drug
* Professional or ancillary personnel involved with this study

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2005-07; Primary Completion 2007-10 (Actual); Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events | One month

SECONDARY OUTCOMES:
Changes in oxygenation, perfusion and cardiovascular status | 3 days
Number and type of cardiac rhythm disturbances | 3 days
Number and duration of intraoperative hypotensive episodes | 6 hours
Incidence of pharmacologic interventions for cardiovascular support | 3 days
Duration of supplemental oxygen use | 3 days
Volume of intravenous fluid administered | 3 days
Blood products administered | 3 days

CONTACTS AND LOCATIONS:
Overall Officials: John Ulatowski, M.D., Ph.D., Principal Investigator — Johns Hopkins University; Peter E. Keipert, Ph.D., Study Director — Sangart, Inc.
Locations (1):
- Johns Hopkins Medical Institutions, Baltimore, Maryland, United States

REFERENCES:
- [Background] Bjorkholm M, Fagrell B, Przybelski R, Winslow N, Young M, Winslow RM. A phase I single blind clinical trial of a new oxygen transport agent (MP4), human hemoglobin modified with maleimide-activated polyethylene glycol. Haematologica. 2005 Apr;90(4):505-15. PMID 15820947
- [Background] Young MA, Riddez L, Kjellstrom BT, Bursell J, Winslow F, Lohman J, Winslow RM. MalPEG-hemoglobin (MP4) improves hemodynamics, acid-base status, and survival after uncontrolled hemorrhage in anesthetized swine. Crit Care Med. 2005 Aug;33(8):1794-804. doi: 10.1097/01.ccm.0000172648.55309.13. PMID 16096458
- [Background] Tsai AG, Cabrales P, Manjula BN, Acharya SA, Winslow RM, Intaglietta M. Dissociation of local nitric oxide concentration and vasoconstriction in the presence of cell-free hemoglobin oxygen carriers. Blood. 2006 Nov 15;108(10):3603-10. doi: 10.1182/blood-2006-02-005272. Epub 2006 Jul 20. PMID 16857991
- [Background] Winslow RM. Current status of oxygen carriers ('blood substitutes'): 2006. Vox Sang. 2006 Aug;91(2):102-10. doi: 10.1111/j.1423-0410.2006.00789.x. PMID 16907870
- [Background] Olofsson C, Ahl T, Johansson T, Larsson S, Nellgard P, Ponzer S, Fagrell B, Przybelski R, Keipert P, Winslow N, Winslow RM. A multicenter clinical study of the safety and activity of maleimide-polyethylene glycol-modified Hemoglobin (Hemospan) in patients undergoing major orthopedic surgery. Anesthesiology. 2006 Dec;105(6):1153-63. doi: 10.1097/00000542-200612000-00015. PMID 17122578
- [Background] Winslow RM. Red cell substitutes. Semin Hematol. 2007 Jan;44(1):51-9. doi: 10.1053/j.seminhematol.2006.09.013. PMID 17198847
- See also: Click here for more information about Sangart, Inc. — http://www.sangart.com